CLINICAL TRIAL: NCT05466877
Title: Phase II Clinical Trial of Safety, Pharmacokinetics and Preliminary Efficacy of MG-K10 Humanized Monoclonal Antibody Injection in Adult Atopic Dermatitis
Brief Title: A Study of MG-K10 in Subjects With Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-K10-AD-2
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: A Phase II Study of the Safety, Pharmacokinetics, Dose-Ranging and Preliminary Efficacy of MG-K10 Humanized Monoclonal Antibody Injection in Adult Patients with Moderate-to-Severe Atopic Dermatitis
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MG-K10 Regimen 1 (Experimental): subcutaneous injection every 4 weeks (placebo injections at 2, 6, 10, 14 weeks to maintain blindness)
  Interventions: Drug: MG-K10
- MG-K10 Regimen 2 (Experimental): subcutaneous injection every 2 weeks
  Interventions: Drug: MG-K10
- MG-K10 Regimen 3 (Experimental): subcutaneous injection every 4 weeks (placebo injections at 2, 6, 10, 14 weeks to maintain blindness)
  Interventions: Drug: MG-K10
- Placebo (Placebo Comparator): subcutaneous injection every 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MG-K10 — MG-K10 Humanized Monoclonal Antibody Injection
  Arms: MG-K10 Regimen 1; MG-K10 Regimen 2; MG-K10 Regimen 3
Drug: Placebo — MG-K10 Humanized Monoclonal Antibody Injection
  Arms: Placebo

SUMMARY:
This study evaluates the preliminary efficacy of MG-K10 in subjects with moderate to severe asthma, and provides a basis for the design and dosing regimen of phase III clinical trials.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled Phase II study. It is planned to enroll approximately 160 adult patients with moderate-to-severe AD uncontrolled by topical therapy, who will receive multiple subcutaneous injections. The study was divided into a screening period (1-5 weeks), a treatment period (16 weeks), and a safety follow-up (8 weeks).

ELIGIBILITY:
key Inclusion Criteria:

1. Aged 18 - 70 years (inclusive), male or female;
2. Patients diagnosed with AD according to American Academy of Dermatology Consensus Criteria (2014) for at least 6 months prior to screening and meet the following criteria:

   * EASI score ≥ 16 at the screening and baseline visits;
   * IGA score ≥ 3 at the screening and baseline visits;
   * AD affected body surface area (BSA) percent ≥10% at the screening and baseline visits;
   * Documented recent history (within 6 months before the screening) of inadequate response to treatment with potent topical corticosteroids for at least 4 weeks or super-potent topical corticosteroids for at least 2 weeks, or topical calcineurin inhibitors for 4 weeks, or prior systemic use of corticosteroids or immunosuppressive agents for more than 2 weeks;

Key Exclusion Criteria:

1. Subjects currently diagnosed with other active skin disorders (e.g., psoriasis or lupus erythematosus) that may affect AD evaluation;
2. Subjects with concomitant diseases that may require systemic hormone therapy or other interventions or require active and frequent monitoring;
3. Subjects with unstable or not well controlled apparent cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological and psychological diseases that is considered by the investigator to be clinically significant；
4. Patients with ocular diseases that are not suitable for enrollment by the investigator；
5. Use of biological agents within 12 weeks prior to randomization or within 5 half-lives (whichever is longer)；
6. Use of topical corticosteroids, topical calcineurin inhibitors, antibiotic compound cream and other topical products for AD treatment within 1 week prior to randomization;
7. chest X-ray or CT examination within 3 months prior to screening/during the screening period suggests the presence of active tuberculosis infection；
8. History of parasitic infection or travel to endemic areas (South America and Africa) half a year prior to screening。

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2024-05-26 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in EASI | 16 weeks
  Percentage change from baseline in eczema area and severity index (EASI) score

SECONDARY OUTCOMES:
Proportions of subjects achieving EASI-75 | 16 weeks
  Proportions of subjects achieving EASI-75 (≥ 75% decrease from baseline in EASI score) at W16
Proportions of subjects achieving IGA score of 0/1 point and a decrease of ≥ 2 points from baseline | 2, 4, 8, 12, 16, 20 ,24 weeks
  Proportions of subjects achieving IGA score of 0/1 point and a decrease of ≥ 2 points from baseline
The change in NRS weekly | 2, 4, 8, 12, 16, 20 ,24 weeks
  The change in NRS weekly mean score and percentage change from baseline at W2, W4, W8, W12, W16, W20, and W24
Percentage change from baseline in EASI score | 2, 4, 8, 12, 20 ,24 weeks
  Percentage change from baseline in EASI score at Weeks W2, W4, W8, W12, W20, and W24
Proportions of subjects achieving EASI-50 | 2, 4, 8, 12, 16, 20 ,24 weeks
  Proportions of subjects achieving EASI-50 (≥ 50% decrease in EASI score from baseline) at W2, W4, W8, W12, W16, W20, and W24
Proportions of subjects achieving EASI-75 | 2, 4, 8, 12, 20 ,24 weeks
  Proportions of subjects achieving EASI-75 at W2, W4, W8, W12, W20, and W24
Proportions of subjects achieving EASI-90 | 2, 4, 8, 12, 16, 20 ,24 weeks
  Proportions of subjects achieving EASI-90 (≥ 90% decrease in EASI score from baseline) at W2, W4, W8, W12, W16, W20, and W24
Absolute change from baseline in EASI scores | 2, 4, 8, 12, 16, 20 ,24 weeks
  Absolute change from baseline in EASI scores at W2, W4, W8, W12, W16, W20, and W24
Absolute and percentage change from baseline in BSA score of Atopic Dermatitis | 2, 4, 8, 12, 16, 20 ,24 weeks
  Absolute and percentage change from baseline in BSA score of Atopic Dermatitis at W2, W4, W8, W12, W16, W20, and W24
Proportions of subjects with a decrease in IGA score from baseline of ≥ 2 | 2, 4, 8, 12, 16, 20 ,24 weeks
  Proportions of subjects with a decrease in IGA score from baseline of ≥ 2 at W2, W4, W8, W12, W16, W20 and W24
Proportions of subjects with a decrease in IGA score from baseline of ≥ 3 | 2, 4, 8, 12, 16, 20 ,24 weeks
  Proportions of subjects with a decrease in IGA score from baseline of ≥ 3 at W2, W4, W8, W12, W16, W20 and W24
Absolute change in POEM from baseline | 2, 4, 8, 12, 16, 20 ,24 weeks
  Absolute change in patient oriented eczema measure (POEM) from baseline at W2, W4, W8, W12, W16, W20 and W24
Absolute change in DLQI score from baseline | 2, 4, 8, 12, 16, 20 ,24 weeks
  Absolute change in dermatology life quality index (DLQI) score from baseline at W2, W4, W8, W12, W16, W20 and W24
Pharmacokinetic concentration | 24 weeks
  To evaluate the Pharmacokinetic concentration of MG-K10
thymus activation regulated chemokine (TARC) | 24 weeks
  At each evaluation time point, the changes of thymus activation regulated chemokine (TARC) were compared with baseline
serum immunoglobulin E (IgE) | 24 weeks
  At each evaluation time point, the changes of serum immunoglobulin E (IgE)were compared with baseline
Incidence of Adverse events (AEs) | 24 weeks
  Including vital signs, physical examinations, laboratory tests, and 12-lead electrocardiograms (ECGs)
Anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs) | 24 weeks
  Incidence of anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs) (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Xu, Medical Ph.D, Principal Investigator — Huashan Hospital
Locations (2):
- China (2):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Huashan Hospital Affiliated to Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No